CLINICAL TRIAL: NCT04190212
Title: Examining the Role of High-intensity Interval Training on Glucose Variability and Symptomatology: A Novel Approach for Patients With Atrial Fibrillation and Diabetes
Brief Title: The Effect of High-Intensity Interval Training on Glucose Variability and Atrial Fibrillation Symptoms
Acronym: Glucose-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 20190687
Record Dates: First submitted 2019-11-29; First posted 2019-12-09 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation; Type 2 Diabetes
Keywords: high-intensity interval training; glycemic variability; continuous glucose monitoring system
MeSH Terms: conditions — Atrial Fibrillation; Diabetes Mellitus, Type 2 | interventions — High-Intensity Interval Training; Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity interval training (Experimental): Participants will complete 12 supervised high-intensity interval exercise sessions (3 times weekly for 4 weeks).
  Interventions: Behavioral: High-intensity interval training + standard care
- Standard care (No Intervention): Participants will not participate in on-site supervised exercise sessions.

INTERVENTIONS:
Behavioral: High-intensity interval training + standard care — HIIT sessions will include: (1) warm-up for 2 minutes at 50% of peak power output (PPO); (2) 2 x 8-minute interval training blocks (total: 16 minutes) of 30-seconds at 80-100% of PPO interspersed with 30-seconds active recovery, 4 minutes of recovery will be permitted between the blocks; and, (3) 2 minute cool-down at 25% of PPO after the last 30-second exercise bout.
  Arms: High-intensity interval training

SUMMARY:
The incidence of atrial fibrillation (AF), the most common heart rhythm disorder, is increasing. The symptoms of AF include: unpleasant heartbeats; difficulty breathing; tiredness; dizziness; and, reduced exercise capacity. Patients with AF have lower quality of life, higher mental distress, and higher risk of heart disease and stroke when compared to the general population. Further, patients with non-permanent AF tend to experience more severe symptoms and substantial reductions in quality of life when compared to patients with permanent AF.

Type 2 diabetes increases the risk of developing AF and accounts for about 20% of patients with non-permanent AF. High blood glucose concentrations and increased blood glucose fluctuations (large and frequent upward and downward blood glucose swings) are commonly seen in type 2 diabetes. Increased blood glucose fluctuations may worsen AF symptoms and quality of life in patients with AF.

Exercise improves quality of life and mental health and reduces risk of developing heart disease and stroke. However, no clinical guidelines for managing AF include exercise. High-intensity interval training (HIIT), a form of exercise that alternates between intense bouts of exercise and less intense recovery periods, is a time-efficient approach to improve blood glucose fluctuations in type 2 diabetes. In healthy individuals and in patients with coronary artery disease, HIIT also improves quality of life and mental health. Currently, the effect of HIIT on blood glucose fluctuations, AF symptom severity and quality of life in patients with AF living with type 2 diabetes is unknown. Also, the links between blood glucose fluctuations and AF symptom severity and quality of life have not been investigated.

DETAILED DESCRIPTION:
There is a global epidemic of AF, the most common sustained cardiac arrhythmia, and type 2 diabetes (T2D). Given an aging population and physically inactive lifestyles, the prevalence of AF and T2D is expected to increase. AF is a progressive disorder with three principal subtypes: paroxysmal AF (AF that self-terminates within <7 days), persistent AF (AF that lasts >7 days and is terminated by medications or procedures) and permanent AF (patient and treating physician agree not to pursue further intervention). AF-related symptoms are disabling and highly variable, including exercise intolerance, palpitations, breathlessness, fatigue, dizziness and mental distress. Patients with non-permanent AF experience more severe symptoms when compared to those with permanent AF, and suffer from substantial reductions in quality of life (QoL) and increased risk of major cerebrovascular events, cardiovascular events and mortality.

T2D is a risk factor for developing AF and approximately 20% of non-permanent AF patients (i.e. paroxysmal and persistent AF) suffer from this condition. T2D is characterized by insulin resistance and insulin insufficiency leading to high blood glucose concentrations. Inadequate or poor glycemic control leads to increases in glycemic variability (GV, amplitude and frequency of blood glucose oscillations from either high to low or low to high). GV is considered to exacerbate AF symptoms severity by increasing: (1) inflammation; (2) oxidative stress; and, (3) autonomic nervous system dysfunction. Emerging evidence also highlights associations between GV and poor QoL and negative mood in patients with T2D.

High-intensity interval training (HIIT), a form of exercise that involves periods of short, intense exercise bouts interspersed by less intense recovery periods, has emerged as a time-efficient and practical approach to improving GV. Importantly, only 10 HIIT sessions over 2 weeks have been shown to lower GV in patients with T2D. A systematic review (N=50 studies) revealed that HIIT improves insulin resistance and blood glucose control (glycated hemoglobin A1C) when compared to controls (i.e. no exercise) in patients with metabolic syndrome or T2D. HIIT also increases QoL in patients with coronary artery disease (CAD) following 4 weeks of exercise training; reduces inflammatory markers (i.e. interleukin-6 [IL-6] and C-reactive protein [CRP]30) in patients with CAD; attenuates markers of oxidative stress in healthy adults in 3 weeks; and improves cardiac autonomic nervous system function in healthy sedentary men in 2 weeks.

The recent American Diabetes Association guidelines recommend HIIT as a strategy to control blood glucose in patients with T2D. However, neither national nor international clinical guidelines for managing AF include exercise. The absence of exercise from these guidelines in the face of increasing evidence of its physical and mental health benefits reflects a lost opportunity to provide AF patients with better treatment options, particularly those who suffer from concomitant T2D. The effects of HIIT on GV, AF symptom severity and QoL in non-permanent AF patients with T2D are unknown, and the associations between GV and AF symptom severity and QoL remain to be investigated. Examining the impact of HIIT on GV, AF symptom severity and QoL may provide a novel, feasible and time-efficient therapeutic option for non-permanent AF patients with T2D who are searching for better treatment options.

ELIGIBILITY:
Inclusion Criteria:

* non-permanent atrial fibrillation
* diagnosed with type 2 diabetes
* non-smokers
* able to perform a symptom-limited cardiopulmonary exercise test (CPET)
* rate controlled with a resting ventricular rate of ≤110 beats per minute

Exclusion Criteria:

* uncontrolled type 2 diabetes (A1C >10 % or presence of type 2 diabetes-related complications
* on exogenous insulin
* unstable diagnosed angina
* diagnosed severe mitral or aortic stenosis
* diagnosed hypertrophic obstructive cardiomyopathy with significant obstruction
* presence of self-reported alcohol or substance abuse
* unable to provide written, informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Glucose variability | From baseline to follow-up after 4-week intervention
  Change in glucose variability as measured by the continuous glucose monitoring system

SECONDARY OUTCOMES:
Atrial fibrillation symptom severity | From baseline to follow-up after 4-week intervention
  Changes in atrial fibrillation symptom severity as assessed by the University of Toronto Atrial Fibrillation Severity Scale (AFSS). The questions include: AF frequency; overall severity; duration of AF episodes; frequency of hospitalization, visits to emergency room and specialist; and overall well-being (Likert scale with 1 indicating "worst possible life" to 10 indicating "best possible life").
Atrial fibrillation-related quality of life | From baseline to follow-up after 4-week intervention
  Change in the AF-related quality of life will be assessed by the Atrial Fibrillation Effect on Quality of Life (AFEQT) Questionnaire.The questionnaire includes Likert scale ranging from 1 to 7. The score will be transformed to a 0 to 100 scale where higher score represents better AF-related quality of life.
General quality of life | From baseline to follow-up after 4-week intervention
  Change in general quality of life will be assessed by the Short Form 36 Health Survey Questionnaire (SF-36). It yields an 8-scale profile of functional health and well-being scores, with higher scores indicating better quality of life.
Sleep quality | From baseline to follow-up after 4-week intervention
  Change in the sleep quality will be assessed by the 3-day sleep diary and Pittsburgh Sleep Quality index (PSQI). A global PSQI score ranges from 0 to 21 with higher scores indicating worse sleep quality.
Changes in blood biomarker concentrations | From baseline to follow-up after 4-week intervention
  Changes in the blood biomarker concentrations linked to glucose variability and AF symptom severity.

OTHER OUTCOMES:
Link between glucose variability and atrial fibrillation symptom severity | From baseline to follow-up after 4-week intervention
  Correlation between glucose variability and atrial fibrillation symptom severity measured by the University of Toronto Atrial Fibrillation Severity Scale (AFSS)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Reed, PhD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada